CLINICAL TRIAL: NCT00057005
Title: Phase I Study of Anti-Human CD45 Monoclonal Antibodies in Patients With Advanced Leukemia Prior to Allogeneic Stem Cell Transplantation (ADVL)
Brief Title: Anti-Human CD45 Monoclonal Antibodies in Patients With Advanced Leukemia Prior to Allogeneic Stem Cell Transplantation
Acronym: ADVL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Pediatrics-Hem-Onc Cell & Gene, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12870; ADVL; NCT00601380 (obsolete NCT alias)
Record Dates: First submitted 2003-03-26; First posted 2003-03-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: LEUKEMIA
Keywords: LEUKEMIA
MeSH Terms: conditions — Leukemia | interventions — Alemtuzumab; Cytarabine; Cyclophosphamide; Mesna; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CAMPATH-1H; Drug: Anti-CD45; Drug: Ara-C; Drug: Cyclophosphamide; Drug: Mesna; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: CAMPATH-1H — Day-8 through Day-6 according to institutional SOPs
Drug: Anti-CD45 — Day-5 400 μg/kg
Drug: Ara-C — day-7 through day-5 3000 mg/m2 q 12h
Drug: Cyclophosphamide — Day-7 through Day-6 45 mg/kg
Drug: Mesna — Days -7 and -6 45 mg/kg divided into 5 doses
Radiation: Total Body Irradiation — 150 cGy x 2 (5/6 matched related) 180 cGy x 2 (5/6 matched unrelated)

SUMMARY:
Participants in this study have a hematologic malignancy which is a disorder in the bone marrow that affects the body's ability to create blood. Participants might benefit from receiving an allogeneic stem cell transplant (meaning the cells come from a donor). The participants donor is a family member. Stem cells are cells in the bone marrow and blood that can form a whole new blood system.

DETAILED DESCRIPTION:
Patients are given high doses of chemotherapy before receiving a stem cell transplant to keep their immune system from rejecting the donor stem cells and to kill any diseased cells that remain in the body. To try and improve on the results of transplants that use high dose chemotherapy alone, we are adding an agent called anti-CD45 to the treatment prior to the stem cell transplant. Anti-CD45 is an antibody that specifically finds and destroys leukemia cells.

Patients will receive the anti-CD45 with high dose chemotherapy (including Ara-C and Cyclophosphamide) and radiotherapy. Patients will also receive Mesna which is a drug that helps prevent bladder damage which can be caused by the cyclophosphamide. High dose radiotherapy is also known as Total Body Irradiation or TBI.

Patients will receive the anti-CD45, high dose chemotherapy, and high dose radiotherapy before the stem cell transplant. We expect participation in this study will last 2 years.

A summary of the treatment follows:

* Day - 7: Ara-C, Cyclophosphamide, Mesna
* Day - 6: Ara-C, Cyclophosphamide, Mesna
* Day - 5: Ara-C, Anti-CD45
* Day - 4: Anti-CD45, TBI
* Day - 3: Anti-CD45, TBI
* Day - 2: Anti-CD45, TBI
* Day - 1: TBI
* Day 0: Stem Cell Infusion (transplant)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced leukemia or other hematologic malignancy including AML, ALL, CML, and MDS. Advanced features include: a) Induction failure, prolonged induction beyond 6 weeks b) Incomplete response to salvage therapy c) CML in blast crisis or acute leukemia in chemotherapy resistant relapse d) secondary leukemia or secondary myelodysplastic disease
2. Patients must have a suitable HLA identical sibling donor or 5/6 matched related donor, or fully matched or 5/6 matched unrelated donor, or haploidentical related donor.

Exclusion Criteria:

1. Patients with a life expectancy (2X normal for age) 7. Patients with known allergy to rat serum products 8. Patients with a Lansky score <60% or Karnofsky score <60%. 9. Patients with severe infection that on evaluation by the PI precludes ablative radio/chemotherapy or successful transplantation. 10. Patients with sever personality disorder or mental illness. 11. Patients with documented HIV positivity 12. Pregnant or lactating females

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2003-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the toxicity and the anti-tumor activity of anti-human CD45 antibodies (anti-CD45) administered to patients with relapsed/resistant leukemia prior to bone marrow transplantation. | 28 days and 100 days post transplant

SECONDARY OUTCOMES:
To describe the effects of anti-CD45 on normal hematopoiesis and on complement levels and to describe the effects of anti-CD45 on leukemic blast cells. | 100 days post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MD, Study Chair — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas